CLINICAL TRIAL: NCT03678038
Title: Comparing the Efficacy of Rotator Interval Steroid Injection Versus Steroid Intraarticular Hydrodilatation in the Treatment of Frozen Shoulder
Brief Title: Comparison of Rotator Interval Injection Versus Intraarticular Hydrodilatation in Frozen Shoulder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-07-008B
Record Dates: First submitted 2018-09-09; First posted 2018-09-19 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Adhesive Capsulitis
Keywords: adhesive capsulitis
MeSH Terms: conditions — Bursitis | interventions — Triamcinolone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rotator interval injection (Experimental): patient received ultrasound-guided steroid injection via rotator interval
  Interventions: Drug: Triamcinolone (Shincort) injection to rotator interval
- posterior recess injection (Active Comparator): patient received ultrasound-guided steroid injection via posterior recess
  Interventions: Drug: Triamcinolone (Shincort) injection to posterior glenuhumeral recess

INTERVENTIONS:
Drug: Triamcinolone (Shincort) injection to rotator interval — via rotator interval.
  Arms: rotator interval injection
Drug: Triamcinolone (Shincort) injection to posterior glenuhumeral recess — via posterior glenuhumeral recess
  Arms: posterior recess injection

SUMMARY:
This study was conducted to compare the efficacy of hydrodilatation with steroid via posterior approach versus rotator interval approach for treating patients with adhesive capsulitis.

DETAILED DESCRIPTION:
Adhesive capsulitis is a common cause of shoulder pain, and the efficacy of most interventions is limited. This study was conducted to compare the efficacy of rotator interval injection with steroid with that of steroid hydrodilatatoin for treating adhesive capsulitis.

Design: a prospective, single-blinded, randomized, clinical trial

Patient and methods:

Patients with adhesive capsulitis were enrolled and randomly allocated into group 1 ( ultrasound guided rotator interval injection ) and group 2 (ultrasound guided steroid hydrodilatation). The patients were evaluated before treatment and were reevaluated 0, 6, and 12 weeks after the beginning of the treatment. Outcomes measures included a pain scale (visual analog scale), range of motion, Constant shoulder score, and Shoulder Pain And Disability Index.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of frozen shoulder by physical examination and ultrasonography

Exclusion Criteria:

1. other conditions involving the shoulder ( rheumatoid arthritis, Hill-Sachs lesions,osteoporosis, or malignancies in the shoulder region)
2. neurologic deficits affecting shoulder function in normal daily activities
3. shoulder pain caused by cervical radiculopathy
4. a history of drug allergy to xylocaine or corticosteroid
5. pregnancy or lactation;
6. received injection into the affected shoulder during the preceding 3 months
7. history of surgeries on the affected shoulders
8. Secondary frozen shoulder

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Shoulder Pain And disability index | Change of the score between 6 weeks and baseline, and change of the score between 12 weeks and baseline
  The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. The pain dimension consists of five questions regarding the severity of an individual's pain. Functional activities are assessed with eight questions designed to measure the degree of difficulty an individual has with various activities of daily living that require upper-extremity use. The SPADI takes 5 to 10 minutes for a patient to complete and is the only reliable and valid region-specific measure for the shoulder.function. The score is divided into four sections: pain, activity of daily living, ROM and strength

SECONDARY OUTCOMES:
pain intensity | Change of the score between 6 weeks and baseline, and change of the score between 12 weeks and baseline
  pain intensity was measured by visual analog scale. Each patient was asked to indicate his/her current level of pain by marking a point on a 100-mm VAS, for which 0 represented no pain and 100 represented unbearable pain.
glenohumeral joint range of motion | Change at baseline, 6 weeks, 12 weeks
  Shoulder flexion, abduction, external rotation and internal rotation were measured with goniometer with patient in supine position

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No